CLINICAL TRIAL: NCT03879733
Title: THRIVE BY 3 Preventive Knowledge Enhancement & Tailored Quality-building in Daycare to Promote Development/ Mental Health in 1&2 Year-olds
Brief Title: THRIVE BY 3 Daycare to Promote Development/ Mental Health in 1&2 Year-olds
Acronym: Tb3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: Norwegian University of Science and Technology (Other); BI Norwegian Business School - Oslo campus (Unknown); University of Washington (Other); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Elisabet Solheim Buøen, Clinical psychologist, PhD, Regionsenter for barn og unges psykiske helse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 260624
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Childcare Quality; Child Development
Keywords: childcare; quality; universal prevention; mental health; well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participating childcare centers are randomized to either a wait list control- group or an intervention group. The wait-list control group will receive the intervention after 1 year.
Who Masked: Participant
Masking Description: The participating child-care centers, staff, parents and children are blind to the study conditions prior to consenting. After randomization the participants know if they get the intervention or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The group of childcare centers that will receive the intervention during 10 months from sept 2018 - June 2019
  Interventions: Behavioral: Thrive by Three
- Wait-list control (Other): Will receive no intervention and continue with business as usual during the primary intervention period Sept. 2018 - June 2019.
  Will receive the intervention from Sept. 2019 - June 2020.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Thrive by Three — The intervention consists of the following components:
  1. Measurement of daycare quality with CLASS (Classroom Assessment Scoring System) 3 times during the intervention period
  2. Feedback to group staff on 8 CLASS-quality dimensions
  3. Monthly supervision of staff on two levels: supervision of daycare staff, and supervision of supervisors
  4. Competence building with all staff: 3 full training days, plus 2 extra training days for pedagogical leaders/supervisors
  5. Written material to parents, supervisors, and staff
  6. Web page for staff and parents: tf3.no
  Arms: Intervention group
Behavioral: Treatment as usual (TAU) — The wait-list control group will continue with their daily activities and work in the childcare as usual. The wait list control group will have received general information about the study prior to consenting, however no materials or are provided by project. The child-care centers in the control conditions will receive a gift certificate of 3000 Norwegian Crones (NOK) by the end of the intervention period.
  Arms: Wait-list control

SUMMARY:
This study evaluates a preventive, knowledge enhancement and tailored quality building intervention to promote development and mental health in 1 and 2 year-olds. Half of the participating childcare centers will get the intervention (intervention group) and half will get the intervention after 1 year (waitlist-control).

DETAILED DESCRIPTION:
Mental health problems manifest already in preschool age and continue into middle and late childhood. However, research strongly indicates that mental health problems appear even among 1-2 year olds. Because 80% of Norwegian under 3 years attend childcare, and stay there for long hours, interventions targeting caregiver-child interactions may prove an important avenue towards universal prevention of mental health problems.

Since requirements for high quality is not sufficiently met in many Norwegian childcare centers today, a cost-efficient, sustainable model of intervention is called for to enhance and track the quality of childcare for 1-3 year olds. The investigators in the study will break new grounds by, conducting a cluster randomized control trial of a newly developed comprehensive intervention for promoting mental health among toddlers in childcare, the Thrive by Three. Because, high quality childcare is in a unique position to prevent developmental trajectories leading to mental health problems and to early identify children in need of help, effective quality enhancing interventions will be of great value for the Norwegian society, both on individual, family, community and national level. The primary objective of the project is thus to investigate whether the intervention Thrive by Three will improve childcare quality, and strengthen children's mental health and development. It is hypothesized that the intervention will prove superior to the wait-list control after the 10 month intervention period and at 12 months follow-up with respect to childcare quality and children's mental health, development and well-being. Our secondary objective is to investigate the cost-effectiveness of the intervention and whether effects are moderated by characteristics of the children, caregivers and/or implementation outcomes. In a subsample of approximately 300 children the investigators will sample cortisol at two time points (pre and post intervention) to investigate whether quality enhancement alters the cortisol level in children in childcare, compared to cortisol secretion at home. User perspectives and experience with Thrive by Three will be captured through qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* Children: All children aged 12 months to 36 months attending one of the selected childcare-centers.
* Child care centers: Childcare centers with groups for children aged 12-36 months was selected within each municipality, after the municipalities had consented to participate in the study. Child care centers volunteered to participate in the study.

Exclusion Criteria:

* Children: None
* Child-Care centers: Child care centers in the selected municipalities with only children older than 36 months.

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1531 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Classroom Assessment Scoring System - Toddler (CLASS) (la Paro, M., Hamre, B., & Pianta, R., 2012) | Baseline, 5 months, 10 months and 22 months. Note: not possible at 22 months due to Covid-19
  CLASS is used to measure change in process quality from pre-intervention (baseline) to half way through the intervention (5 months) period, post-intervention (10 months) as well as at 12 months follow up (22 months). CLASS is a multidimensional observational measure of process quality in daycare, for toddlers. Trained observers observe each group of children and staff for 3 loops of 15 minutes. Quality is assessed along 8 dimensions and 2 quality domains. Scores are given on a scale from 1-7 with 7 indicating higher quality, except on the dimension negative climate, where 1 indicates higher quality. The dimension score of negative climate is reversed when domain scores are calculated. Scores of 1-2 indicates low quality, 3-5 mediocre, and 6-7 high. Scores for each cycles are calculated, and averaged to give the dimension scores. Domain scores are then calculated based on the averaged domain scores.
Child Behavior Checklist for preschool children (CBCL)(Achenbach, T. M., 2000) | Baseline, 10 months and 22 months (one year follow up)
  100 item parent report of child behavioral, emotional and social problems. each item is rated as 0 (Not True),1 (Somewhat or Sometimes True), or 2 (Very True, or Often True). Low scores indicate fewer problems. The measure is used to measure change in problem behavior during the intervention period (from baseline to end of intervention), and used as an outcome measure at post intervention (10 months) to see whether children in childcare center where the quality has positively changed during the intervention period will have less problem behavior.
C- Teacher report form for preschool children (C-TRF)(Achenbach, T. M., 2000) | Baseline, 10 months and 22 months (one year follow up)
  100 item teacher report of child behavioral, emotional and social problems. Each item is rated as 0 (Not True),1 (Somewhat or Sometimes True), or 2 (Very True, or Often True). Low scores indicate fewer problems. The measure is used to measure change in problem behavior during the intervention period (from baseline to end of intervention), and used as an outcome measure at post intervention (10 months) to see whether children in childcare center where the quality has positively changed during the intervention period will have less problem behavior.
The Brief Infant-Toddler Social and emotional Assessment (BITSEA) (Briggs-Gowan, M. J., Carter A.S. , Irwin J.R., Wachtel K. & Cicchetti D.V., 2004) | Baseline, 10 months and 22 months (one year follow up)
  BITSEA is a 42 item instrument to assess social-emotional/behavioral problems and delays in social-emotional competence in toddlers. The BITSEA is completed both by parents and child care staff. We use BITSEA to measure change in problem behavior during the intervention period (from baseline to end of intervention), and BITSEA is also used as an outcome measure at post intervention (10 months) and at 12 months follow up (22 months) to see whether children in childcare centers where the quality has positively changed during the intervention period will have less problem behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet S. Buoen, PhD, Principal Investigator — RegionsenterRBUP
Locations (3):
- Norway (3):
  - Regional center for child and adolescent mental health, Eastern and southern Norway, Oslo, Nydalen
  - Norwegian Buisness School, BI, Oslo
  - Norwegian university of Science and Technology (NTNU), Trondheim

REFERENCES:
- [Derived] Buoen ES, Lekhal R, Lydersen S, Berg-Nielsen TS, Drugli MB. Promoting the Quality of Teacher-Toddler Interactions: A Randomized Controlled Trial of "Thrive by Three" In-Service Professional Development in 187 Norwegian Toddler Classrooms. Front Psychol. 2021 Nov 18;12:778777. doi: 10.3389/fpsyg.2021.778777. eCollection 2021. PMID 34867691
- [Derived] Lekhal R, Drugli MB, Berg-Nielsen TS, Buoen ES. A Model of Intervention and Implementation of Quality Building and Quality Control in Childcare Centers to Strengthen the Mental Health and Development of 1-3-Year Olds: Protocol for a Randomized Controlled Trial of Thrive by Three. JMIR Res Protoc. 2020 Oct 13;9(10):e17726. doi: 10.2196/17726. PMID 32773366